CLINICAL TRIAL: NCT00180479
Title: SPIRIT III: A Clinical Evaluation of the Investigational Device XIENCE V® Everolimus Eluting Coronary Stent System (EECSS) in the Treatment of Subjects With de Novo Native Coronary Artery Lesions
Brief Title: SPIRIT III Clinical Trial of the XIENCE V® Everolimus Eluting Coronary Stent System (EECSS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03-360
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2008-12-15 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Stents; Coronary Artery Disease; Total Coronary Occlusion; Coronary Artery Restenosis; Stent Thrombosis; Vascular Disease; Myocardial Ischemia; Coronary Artery Stenosis
Keywords: Everolimus
MeSH Terms: conditions — Coronary Artery Disease; Coronary Restenosis; Vascular Diseases; Myocardial Ischemia; Coronary Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): XIENCE V® Everolimus Eluting Coronary Stent System
  Interventions: Device: XIENCE V® Everolimus Eluting Coronary Stent
- 2 (Active Comparator): TAXUS® EXPRESS2™Paclitaxel Eluting Coronary Stent System
  Interventions: Device: TAXUS® EXPRESS2™ Paclitaxel Eluting Coronary Stent

INTERVENTIONS:
Device: XIENCE V® Everolimus Eluting Coronary Stent — Drug eluting stent implantation stent in the treatment of coronary artery disease.
  Other Names: XIENCE V® Everolimus Eluting Coronary Stent System
  Arms: 1
Device: TAXUS® EXPRESS2™ Paclitaxel Eluting Coronary Stent — Drug eluting stent implantation stent in the treatment of coronary artery disease.
  Other Names: TAXUS® EXPRESS2™ Paclitaxel Eluting Coronary Stent System
  Arms: 2

SUMMARY:
This study is divided into 5 arms:

1. Randomized Clinical Trial (RCT): Prospective, randomized, active-controlled, single blind, parallel two-arm multi-center clinical trial in the United States (US) comparing XIENCE V® Everolimus Eluting Coronary Stent System (CSS) (2.5, 3.0, 3.5 mm diameter stents) to the Food and Drug Administration (FDA) approved commercially available active control TAXUS® EXPRESS2™ Paclitaxel Eluting Coronary Stent (TAXUS® EXPRESS2™ PECS) System
2. US 2.25 mm non-randomized arm using 2.25 mm diameter XIENCE V® Everolimus Eluting CSS
3. US 4.0 mm non-randomized arm using 4.0 mm diameter XIENCE V® Everolimus Eluting CSS
4. US 38 mm non-randomized arm using 38 mm in length XIENCE V® Everolimus Eluting CSS
5. Japanese non-randomized arm using XIENCE V® Everolimus Eluting CSS (2.5, 3.0, 3.5, 4.0 mm diameter stents) in Japan

The TAXUS® EXPRESS2™ Paclitaxel Eluting Coronary Stent System is Manufactured by Boston Scientific.

DETAILED DESCRIPTION:
The purpose of the SPIRIT III clinical trial is to evaluate the safety and efficacy of the XIENCE V® Everolimus Eluting Coronary Stent System (XIENCE V® EECSS). The XIENCE V® EECS (XIENCE V® arm) will be compared to an active control group represented by the FDA approved commercially available Boston Scientific TAXUS® EXPRESS2™ Paclitaxel-Eluting Coronary Stent (TAXUS® EXPRESS2™ PECS) System (TAXUS® arm).

The SPIRIT III clinical trial consists of a randomized clinical trial (RCT) in the US which will enroll approximately 1,002 subjects (2:1 randomization XIENCE V® EECS : TAXUS® EXPRESS2™ PECS) with a maximum of two de novo native coronary artery lesion treatment within vessel sizes >= 2.5 mm and <= 3.75 mm.

The SPIRIT III clinical trial also consists of three concurrent US non-randomized arms (2.25 mm diameter stent, 4.0 mm diameter stent and 38 mm length stent arms) and one Japanese non-randomized arm as follows:

1. 105 subjects with a maximum of two de novo native coronary artery lesion within vessel sizes > 2.25 mm and < 2.5 mm and lesion length <= 22 mm will be enrolled concurrently in the US 2.25 mm non-randomized treatment arm
2. 80 subjects with a maximum of two de novo native coronary artery lesion within vessel sizes > 3.75 mm and >= 4.25 mm and lesion length <= 28 mm will be enrolled concurrently in the US 4.0 mm non-randomized treatment arm
3. 105 subjects with a maximum of two de novo native coronary artery lesion within vessel sizes > 3.0 mm and < 4.25 mm and lesion length > 24 mm and < 32 mm will be enrolled concurrently in the US 38 mm non-randomized treatment arm.
4. 88 Japanese subjects with a maximum of two de novo native coronary artery lesions within vessel sizes >= 2.5 mm and <= 4.25 mm and lesion length <= 28 mm will be enrolled concurrently in the non-randomized Japanese arm.

All subjects in the RCT and the four non-randomized arms will be screened per the protocol required inclusion/exclusion criteria. The data collected will be compared to data from the subjects enrolled into the TAXUS® arm of US RCT.

Subjects enrolled in the US RCT will be sub-grouped based on whether they will have an angiographic and/or an intravascular ultrasound (IVUS) follow-up at 240 days as follows:

Group A: Angiographic and IVUS follow-up at 240 days (N=240) Group B: Angiographic follow-up at 240 days (N=324) Group C: No angiographic or IVUS follow-up (N=438)

All subjects will have clinical follow-up at 30, 180, 240 and 270 days (Data collected through 270 days will be submitted as the primary data set for US and Japanese market approval), and 1, 2, 3, 4, and 5 years (for annual reports).

All subjects enrolled into three US non-randomized arms (N=105 for 2.25 mm arm, N=80 for 4.0 mm arm and N=105 for 38 mm stent arm) will have clinical follow-up at 30, 180, 240, and 270 days, and angiographic follow-up at 240 days. No IVUS follow-up is required for subjects enrolled in these arms.

All subjects enrolled into the Japanese non-randomized arm (N=88) will have clinical follow-up at 30, 180, 240, and 270 days, and angiographic and IVUS follow-up at 240 days.

All subjects who receive a bailout stent will be assigned to Group A follow-up subgroup (angiographic and IVUS follow-up at 240 days after the index procedure), regardless of their primary assignment at randomization. At sites without IVUS capability, subjects receiving bailout stent will be assigned to Group B follow-up subgroup (angiographic follow-up at 240 days after the index procedure). Angiographic follow-up is required for all bailout subjects at 240 days.

Data from the US RCT will be submitted to the FDA as the primary data set for product approval for RVD >= 2.5 mm and <= 3.75 mm (2.5 mm, 3.0 mm and 3.5 mm stents). Combined data of the US trial/Japanese non-randomized arm will be submitted to the Japanese Ministry of Health, Labor and Welfare (MHLW) for Japanese approval for RVD>=2.5 mm and <= 4.25 mm (2.5 mm, 3.0 mm 3.5 mm and 4.0 mm stents). Data from the Japanese non-randomized arm will be submitted to the FDA as additional safety data. Data from the US non-randomized arms of the trial will be the primary data sets for approval for 2.25 mm diameter stent (RVD > 2.25 mm and < 2.5 mm), 4.0 mm diameter stent (RVD > 3.75 mm and <= 4.25 mm) and 38 mm length stent (RVD > 3.0 mm and <= 4.25 mm and lesion length > 24 mm and <= 32 mm), respectively in the US.

A pharmacokinetic substudy will be carried out in a minimum of 5 pre-determined sites in the US and a minimum of 5 pre-determined sites in Japan. In the US, the pharmacokinetics (PK) of everolimus, as delivered by the XIENCE V® EECS will be analyzed in a subset of 15 subjects (minimum) with single vessel/lesion treatment, and up to 20 subjects with dual vessel/lesion treatment, respectively. In Japan, a minimum of 10 subjects with single vessel/lesion treatment and up to 20 subjects with dual vessel/lesion treatment will have a PK measurements performed. These subsets will include subjects receiving overlapping stents.

ELIGIBILITY:
Inclusion Criteria:

* Target lesion(s) must be located in a native epicardial vessel with visually estimated diameter between >= 2.25 mm and <= 4.25 mm and a lesion length <= 32 mm
* The target lesion(s) must be in a major artery or branch with a visually estimated stenosis of >= 50% and < 100% with a thrombolysis in myocardial infarction (TIMI) flow of >= 1
* Non-study, percutaneous intervention for lesions in a non-target vessel is allowed if done >= 90 days prior to the index procedure (subjects who received brachytherapy will be excluded from the trial)

Exclusion Criteria:

* Located within an arterial or saphenous vein graft or distal to a diseased (vessel irregularity per angiogram and > 20% stenosed lesion by visual estimation) arterial or saphenous vein graft
* Lesion involving a bifurcation >= 2 mm in diameter or ostial lesion > 50% stenosed by visual estimation or side branch requiring predilatation
* Located in a major epicardial vessel that has been previously treated with brachytherapy
* Located in a major epicardial vessel that has been previously treated with percutaneous intervention < 9 months prior to index procedure
* Total occlusion (TIMI flow 0), prior to wire passing
* The target vessel contains thrombus
* Another significant lesion (> 40% diameter stenosis [DS]) is located in the same epicardial vessel as the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1002 (Actual)
Dates: Start 2005-06; Primary Completion 2006-12 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg W Stone, MD, Principal Investigator — Columbia University
Locations (65):
- United States (65):
  - Baptist Medical Center Princeton, Birmingham, Alabama
  - Baptist Health System - Montclair, Birmingham, Alabama
  - Arizona Heart Hospital, Phoenix, Arizona
  - Scripps Memorial Hospital, La Jolla, California
  - Good Samaritan Hospital, Los Angeles, California
  - Alta Bates Summit Medical Center, Oakland, California
  - Mercy General Hospital, Sacramento, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Holy Cross Medical Center (prev. North Ridge MC), Fort Lauderdale, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - St. John's Hospital, Springfield, Illinois
  - The Heart Center of IN, LLC, Indianapolis, Indiana
  - Jewish Hospital, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Washington Adventist Hospital, Takoma Park, Maryland
  - St. Joseph Medical Center, Towson, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - St John Hospital & Medical Center, Detroit, Michigan
  - Spectrum Health Hospital, Grand Rapids, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - St. Luke's Hospital, Kansas City, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - St. Patrick Hospital, Missoula, Montana
  - Nebraska Heart Hospital, Lincoln, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack Medical Center, Hackensack, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - St. Joseph's Hospital Health Center, Syracuse, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Medical Center, Raleigh, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - EMH Regional Medical Center, Elyria, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Baptist Medical, Inc., Oklahoma City, Oklahoma
  - Sacred Heart Medical Center, Eugene, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Pinnacle Health @ Harrisburg Hospital, Harrisburg, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Heart Hospital of Austin, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Methodist Hospital, Houston, Texas
  - TexSan Heart Hospital, San Antonio, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Swedish Medical Center, Seattle, Washington
  - St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Result] Stone GW, Midei M, Newman W, Sanz M, Hermiller JB, Williams J, Farhat N, Mahaffey KW, Cutlip DE, Fitzgerald PJ, Sood P, Su X, Lansky AJ; SPIRIT III Investigators. Comparison of an everolimus-eluting stent and a paclitaxel-eluting stent in patients with coronary artery disease: a randomized trial. JAMA. 2008 Apr 23;299(16):1903-13. doi: 10.1001/jama.299.16.1903. PMID 18430909
- [Result] Stone GW, Midei M, Newman W, Sanz M, Hermiller JB, Williams J, Farhat N, Caputo R, Xenopoulos N, Applegate R, Gordon P, White RM, Sudhir K, Cutlip DE, Petersen JL; SPIRIT III Investigators. Randomized comparison of everolimus-eluting and paclitaxel-eluting stents: two-year clinical follow-up from the Clinical Evaluation of the Xience V Everolimus Eluting Coronary Stent System in the Treatment of Patients with de novo Native Coronary Artery Lesions (SPIRIT) III trial. Circulation. 2009 Feb 10;119(5):680-6. doi: 10.1161/CIRCULATIONAHA.108.803528. Epub 2009 Jan 26. PMID 19171853
- [Result] Lansky AJ, Ng VG, Mutlu H, Cristea E, Guiran JB, Midei M, Newman W, Sanz M, Sood P, Doostzadeh J, Su X, White R, Cao S, Sudhir K, Stone GW. Gender-based evaluation of the XIENCE V everolimus-eluting coronary stent system: clinical and angiographic results from the SPIRIT III randomized trial. Catheter Cardiovasc Interv. 2009 Nov 1;74(5):719-27. doi: 10.1002/ccd.22067. PMID 19530147
- [Derived] Genereux P, Rutledge DR, Palmerini T, Caixeta A, Kedhi E, Hermiller JB, Wang J, Krucoff MW, Jones-McMeans J, Sudhir K, Simonton CA, Serruys PW, Stone GW. Stent Thrombosis and Dual Antiplatelet Therapy Interruption With Everolimus-Eluting Stents: Insights From the Xience V Coronary Stent System Trials. Circ Cardiovasc Interv. 2015 May;8(5):e001362. doi: 10.1161/CIRCINTERVENTIONS.114.001362. PMID 25940520
- [Derived] Muramatsu T, Onuma Y, van Geuns RJ, Chevalier B, Patel TM, Seth A, Diletti R, Garcia-Garcia HM, Dorange CC, Veldhof S, Cheong WF, Ozaki Y, Whitbourn R, Bartorelli A, Stone GW, Abizaid A, Serruys PW; ABSORB Cohort B Investigators; ABSORB EXTEND Investigators; SPIRIT FIRST Investigators; SPIRIT II Investigators; SPIRIT III Investigators; SPIRIT IV Investigators. 1-year clinical outcomes of diabetic patients treated with everolimus-eluting bioresorbable vascular scaffolds: a pooled analysis of the ABSORB and the SPIRIT trials. JACC Cardiovasc Interv. 2014 May;7(5):482-93. doi: 10.1016/j.jcin.2014.01.155. Epub 2014 Apr 16. PMID 24746650
- [Derived] Claessen BE, Smits PC, Kereiakes DJ, Parise H, Fahy M, Kedhi E, Serruys PW, Lansky AJ, Cristea E, Sudhir K, Sood P, Simonton CA, Stone GW. Impact of lesion length and vessel size on clinical outcomes after percutaneous coronary intervention with everolimus- versus paclitaxel-eluting stents pooled analysis from the SPIRIT (Clinical Evaluation of the XIENCE V Everolimus Eluting Coronary Stent System) and COMPARE (Second-generation everolimus-eluting and paclitaxel-eluting stents in real-life practice) Randomized Trials. JACC Cardiovasc Interv. 2011 Nov;4(11):1209-15. doi: 10.1016/j.jcin.2011.07.016. PMID 22115661
- [Derived] Planer D, Smits PC, Kereiakes DJ, Kedhi E, Fahy M, Xu K, Serruys PW, Stone GW. Comparison of everolimus- and paclitaxel-eluting stents in patients with acute and stable coronary syndromes: pooled results from the SPIRIT (A Clinical Evaluation of the XIENCE V Everolimus Eluting Coronary Stent System) and COMPARE (A Trial of Everolimus-Eluting Stents and Paclitaxel-Eluting Stents for Coronary Revascularization in Daily Practice) Trials. JACC Cardiovasc Interv. 2011 Oct;4(10):1104-15. doi: 10.1016/j.jcin.2011.06.018. PMID 22017936
- [Derived] Kereiakes DJ, Sudhir K, Hermiller JB, Gordon PC, Ferguson J, Yaqub M, Sood P, Su X, Yakubov S, Lansky AJ, Stone GW. Comparison of everolimus-eluting and paclitaxel-eluting coronary stents in patients undergoing multilesion and multivessel intervention: the SPIRIT III (A Clinical Evaluation of the Investigational Device XIENCE V Everolimus Eluting Coronary Stent System [EECSS] in the Treatment of Subjects With De Novo Native Coronary Artery Lesions) and SPIRIT IV (Clinical Evaluation of the XIENCE V Everolimus Eluting Coronary Stent System in the Treatment of Subjects With De Novo Native Coronary Artery Lesions) randomized trials. JACC Cardiovasc Interv. 2010 Dec;3(12):1229-39. doi: 10.1016/j.jcin.2010.09.014. PMID 21232716
- [Derived] Caixeta A, Lansky AJ, Serruys PW, Hermiller JB, Ruygrok P, Onuma Y, Gordon P, Yaqub M, Miquel-Hebert K, Veldhof S, Sood P, Su X, Jonnavithula L, Sudhir K, Stone GW; SPIRIT II and III Investigators. Clinical follow-up 3 years after everolimus- and paclitaxel-eluting stents: a pooled analysis from the SPIRIT II (A Clinical Evaluation of the XIENCE V Everolimus Eluting Coronary Stent System in the Treatment of Patients With De Novo Native Coronary Artery Lesions) and SPIRIT III (A Clinical Evaluation of the Investigational Device XIENCE V Everolimus Eluting Coronary Stent System [EECSS] in the Treatment of Subjects With De Novo Native Coronary Artery Lesions) randomized trials. JACC Cardiovasc Interv. 2010 Dec;3(12):1220-8. doi: 10.1016/j.jcin.2010.07.017. PMID 21232715

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1002 subjects were recruited at 65 sites. Eligible subjects invited to participate either in-hospital or in-clinic prior to first procedure and required to provide signed informed consent prior to enrollment. Final eligibility based on angiogram before the intended procedure. Dates of recruitment: 6/22/05 through 3/15/06.
Pre-assignment Details: Subjects were randomized via telephone randomization and stratified by single and dual lesion/vessel treatment, diabetes mellitus status, and study sites. Randomization only occurred after verification of the inclusion/exclusion criteria and successful pre-dilatation. See the Eligibility Criteria (inclusion/exclusion criteria) for details.
Groups:
- XIENCE V® EECSS: XIENCE V® Everolimus Eluting Coronary Stent System
- TAXUS® EXPRESS2™ ECSS: TAXUS® EXPRESS2™ Paclitaxel Eluting Coronary Stent System. 1 patient randomized never signed consent, therefore no data collected. Taxus analysis group = 332.
Period: Overall Study
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Started | 669 | 333 (1 patient randomized never signed consent, therefore no data collected. Analysis group = 332.)
Completed | 653 | 320
Not Completed | 16 | 13
Not completed — Death | 4 | 2
Not completed — Lost to Follow-up | 9 | 7
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Informed consent not signed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS | Total
Number analyzed (Participants) | 669 | 333 | 1002
Age Categorical [Number; unit: participants] — 1 patient randomized never signed consent, therefore no data collected. Taxus analysis group = 332.
  participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 376 | 191 | 567
    >=65 years | 293 | 141 | 434
Age Continuous [Mean (Standard Deviation); unit: years] — 1 patient randomized never signed consent, therefore no data collected. Taxus analysis group = 332.
  years | 63.23 (10.53) | 62.80 (10.24) | 63.08 (10.43)
Gender [Number; unit: participants] — 1 patient randomized never signed consent, therefore no data collected. Taxus analysis group = 332.
  participants
    Female | 200 | 114 | 314
    Male | 469 | 218 | 687
Region of Enrollment [Number; unit: participants] — 1 patient randomized never signed consent, therefore no data collected. Taxus analysis group = 332.
  participants
    United States | 669 | 333 | 1002

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint: In-segment Late Loss (LL)
Description: In-segment minimal lumen diameter (MLD) post-procedure minus (-) in segment MLD at 240 day follow-up and 5 mm proximal and 5mm distal to the stent equals Late Loss. MLD defined: The average of two orthogonal views (when possible) of the narrowest point within the area of assessment.
Time Frame: 240 days
Population: Only a certain number of patients were required to have angiographic follow-up to provide this endpoint information.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 301 | 134
millimeters | 0.14 (0.41) | 0.28 (0.48)
Statistical Analysis 1: Comparison: XIENCE V® EECSS vs TAXUS® EXPRESS2™ ECSS; Primary endpoint analyzed for intent-to-treat & per-treatment evaluable pop. Hypothesis test based on per-subject analysis of intent-to-treat pop. using analysis lesion. The null hypothesis evaluated using non-inferiority test with asymptotic test statistic; Test type: Non-Inferiority or Equivalence — Sample size calculation for endpoint of in-segment LL at 240 days is based on these assumptions: one-tailed non-inferiority= (δ)=0.025, Power=99%, Randomization ratio 2:1, True mean in-seg. LL is assumed to be 0.24 mm in both arms; p < 0.0001, t-test, 1 sided

2. Secondary Outcome: Major Secondary Endpoint: Ischemia Driven Target Vessel Failure (ID-TVF)
Description: The composite endpoint comprised of:
  * Cardiac death (death in which a cardiac cause cannot be excluded)
  * Myocardial infarction (MI, classified as Q-wave and non-Q wave)
  * Ischemia-driven target lesion revascularization (TLR) by CABG or PCI
  * Ischemia-driven target vessel revascularization (TVR) by CABG or PCI
Time Frame: 270 days
Population: All patients in the study underwent clinical follow up to provide the information needed for this endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 657 | 321
percentage of participants | 7.2 | 9.0
Statistical Analysis 1: Comparison: XIENCE V® EECSS vs TAXUS® EXPRESS2™ ECSS; Null hypothesis was evaluated using a non-inferiority Z statistic. Non-inferiority was defined as a one-sided alpha of 0.05 and a difference in TVF rate of no more than 5.5%; Test type: Non-Inferiority or Equivalence — Study had 89% statistical power based on major secondary endpoint to prove non-inferiority of XIENCE® V to TAXUS®, non-inferiority delta=5.5%, true TVF rate 9.4% in both arms with overall 5% alpha (one-sided), assuming 1% subject dropout rate; p < 0.0001, t-test, 1 sided

3. Secondary Outcome: Target Vessel Failure (TVF)
Description: as for outcome 2
Time Frame: 30 days
Population: All patients in the study underwent clinical follow up to provide the information needed for the secondary endpoints. The analysis population at clinical follow-up visits may have changed due to early termination from the study by the patient or physician.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 667 | 330
percentage of participants | 1.6 | 3.3

4. Secondary Outcome: Target Vessel Failure (TVF)
Description: as for outcome 2
Time Frame: 180 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 664 | 326
percentage of participants | 4.1 | 5.5

5. Secondary Outcome: Target Vessel Failure (TVF)
Description: as for outcome 2
Time Frame: 1 year
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 654 | 319
percentage of participants | 8.6 | 11.6

6. Secondary Outcome: Target Vessel Failure (TVF)
Description: as for outcome 2
Time Frame: 2 year
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 637 | 305
percentage of participants | 11.3 | 16.4

7. Secondary Outcome: Target Vessel Failure (TVF)
Description: as for outcome 2
Time Frame: 3 year
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 629 | 305
percentage of participants | 14.3 | 20.0

8. Secondary Outcome: Target Vessel Failure (TVF)
Description: as for outcome 2
Time Frame: 4 year
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 615 | 302
percentage of participants | 18.5 | 22.5

9. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: Revascularization @ target lesion associated w/ any of following:
  (+) functional ischemia study Ischemic symptoms & angiographic diameter stenosis ≥50% by core lab quantitative coronary angiography (QCA) Revascularization of a target lesion w/ angiographic diameter stenosis ≥70% by core laboratory QCA without angina or (+) functional study
Time Frame: 30 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 667 | 330
percentage of participants | 0.4 | 0.3

10. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 9
Time Frame: 180 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 664 | 326
percentage of participants | 1.5 | 2.1

11. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 9
Time Frame: 270 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 659 | 320
percentage of participants | 2.7 | 5.0

12. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 9
Time Frame: 1 years
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 654 | 319
percentage of participants | 3.4 | 5.6

13. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 9
Time Frame: 2 years
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 637 | 305
percentage of participants | 5.7 | 9.2

14. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 9
Time Frame: 3 year
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 629 | 305
percentage of participants | 5.7 | 9.2

15. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 9
Time Frame: 4 year
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 615 | 302
percentage of participants | 8.0 | 10.6

16. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: Revascularization at the target vessel associated with any of the following
  * Positive functional ischemia study
  * Ischemic symptoms and angiographic diameter stenosis ≥ 50% by core laboratory QCA
  * Revascularization of a target vessel with angiographic diameter stenosis ≥ 70% by core laboratory QCA without angina or positive functional study
  Derived from Non-Hierarchical Subject Counts of Adverse Events
Time Frame: 30 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 667 | 330
percentage of participants | 0.3 | 0.9

17. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: as for outcome 16
Time Frame: 180 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 664 | 326
percentage of participants | 1.2 | 1.8

18. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: as for outcome 16
Time Frame: 270 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 659 | 320
percentage of participants | 2.9 | 4.1

19. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: as for outcome 16
Time Frame: 1 year
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 654 | 319
percentage of participants | 3.1 | 4.7

20. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: as for outcome 16
Time Frame: 2 years
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 637 | 305
percentage of participants | 4.9 | 6.6

21. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: as for outcome 16
Time Frame: 3 years
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 629 | 305
percentage of participants | 6.7 | 8.9

22. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: as for outcome 16
Time Frame: 4 years
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 615 | 302
percentage of participants | 7.8 | 9.6

23. Secondary Outcome: Ischemia Driven Major Adverse Cardiac Event (MACE)
Description: The composite endpoint comprised of:
  * Cardiac death
  * Myocardial infarction (MI, classified as Q-wave and non-Q wave)
  * Ischemia-driven target lesion revascularization (TLR) by CABG or PCI
Time Frame: 30 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 667 | 330
percentage of participants | 1.3 | 3.0

24. Secondary Outcome: Ischemia Driven Major Adverse Cardiac Event (MACE)
Description: as for outcome 23
Time Frame: 180 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 664 | 326
percentage of participants | 2.9 | 5.2

25. Secondary Outcome: Ischemia Driven Major Adverse Cardiac Event (MACE)
Description: as for outcome 23
Time Frame: 270 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 659 | 320
percentage of participants | 5.0 | 8.8

26. Secondary Outcome: Ischemia Driven Major Adverse Cardiac Event (MACE)
Description: as for outcome 23
Time Frame: 1 year
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 654 | 319
percentage of participants | 6.0 | 10.3

27. Secondary Outcome: Ischemia Driven Major Adverse Cardiac Event(MACE)
Description: as for outcome 23
Time Frame: 2 years
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 637 | 305
percentage of participants | 7.7 | 13.8

28. Secondary Outcome: Ischemia Driven Major Adverse Cardiac Event (MACE)
Description: as for outcome 23
Time Frame: 3 year
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 629 | 305
percentage of participants | 9.7 | 16.4

29. Secondary Outcome: Ischemia Driven Major Adverse Cardiac Event (MACE)
Description: as for outcome 23
Time Frame: 4 year
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 615 | 302
percentage of participants | 12.8 | 18.5

30. Secondary Outcome: In-stent % Angiographic Binary Restenosis (% ABR) Rate
Description: Percent of subjects with a follow-up in-stent percent diameter stenosis of ≥ 50% per quantitative coronary angiography (QCA)
Time Frame: at 240 days
Population: Only a certain number of patients were required to have angiographic or IVUS follow-up. The analysis population for these follow-ups may have changed due to patient's not completing an angiographic or IVUS follow-up procedure. Patients may also have missed the follow-up visits due to early termination from the study.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 343 | 158
percentage of participants | 2.3 | 5.7

31. Secondary Outcome: In-segment % Angiographic Binary Restenosis (% ABR) Rate
Description: Percent of subjects with a follow-up in-segment percent diameter stenosis of ≥ 50% per QCA
Time Frame: 240 days
Population: as for outcome 30
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 344 | 158
percentage of participants | 4.7 | 8.9

32. Secondary Outcome: Persisting Incomplete Stent Apposition, Late-acquired Incomplete Stent Apposition, Aneurysm, Thrombosis, and Persisting Dissection
Description: Incomplete Apposition (Persisting & Late acquired): Failure to completely appose vessel wall w/ ≥1 strut separated from vessel wall w/ blood behind strut per ultrasound. Aneurysm: Abnormal vessel expansion ≥ 1.5 of reference vessel diameter. Thrombus: Protocol & ARC definition.
  Persisting dissection @ follow-up, present post-procedure.
Time Frame: at 240 days
Population: as for outcome 30
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 90 | 43
percentage of participants | 24.4 | 14.0

33. Secondary Outcome: Acute Success: Clinical Device
Description: Successful delivery and deployment of 1st implanted study stent/s @ the intended target lesion and successful withdrawal of the stent delivery system with final residual stenosis < 50%.
Time Frame: In-hospital
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 763 | 379
percentage of participants | 98.3 | 98.7

34. Secondary Outcome: Acute Success: Clinical Procedure
Description: Successful delivery and deployment of study stent/s @ the intended target lesion and successful withdrawal of the stent delivery system with final residual stenosis < 50%.
Time Frame: In-hospital
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 661 | 331
percentage of participants | 98.5 | 97.3

35. Secondary Outcome: Proximal Late Loss
Description: Proximal Minimum Lumen Diameter (MLD) post-procedure minus proximal MLD at follow-up (proximal defined as within 5 mm of healthy tissue proximal to stent placement)
Time Frame: at 240 days
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 293 | 134
millimeters | 0.12 (0.40) | 0.20 (0.41)

36. Secondary Outcome: Distal Late Loss
Description: Distal MLD post-procedure minus distal MLD at follow-up (distal defined as within 5 mm of healthy tissue distal to stent placement)
Time Frame: 240 days
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 327 | 154
millimeters | 0.09 (0.36) | 0.10 (0.37)

37. Secondary Outcome: In-stent Late Loss
Description: In-stent MLD post-procedure minus in-stent MLD at follow-up (in-stent defined as within the margins of the stent)
Time Frame: at 240 days
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 342 | 158
millimeters | 0.16 (0.41) | 0.30 (0.53)

38. Secondary Outcome: % Volume Obstruction (% VO)
Description: Defined as stent intimal hyperplasia and calculated as 100*(Stent Volume - Lumen Volume)/Stent Volume by IVUS.
Time Frame: at 240 days
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: percent of volume obstruction
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 98 | 39
percent of volume obstruction | 6.91 (6.35) | 11.21 (9.86)

39. Secondary Outcome: In-stent % Diameter Stenosis (% DS)
Description: In-stent: Within the margins of the stent, the value calculated as 100 * (1 - in-stent MLD/RVD) using the mean values from two orthogonal views (when possible) by QCA.
Time Frame: at 240 days
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: percent diameter stenosis
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 343 | 158
percent diameter stenosis | 5.92 (16.40) | 10.30 (21.43)

40. Secondary Outcome: In-segment % Diameter Stenosis (% DS)
Description: Within the margins of the stent, 5 mm proximal and 5 mm distal to the stent, the value calculated as 100 * (1 - in-segment MLD/RVD) using the mean values from two orthogonal views (when possible) by QCA.
Time Frame: 240 days
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: percent of in-segment diameter stenosis
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 344 | 158
percent of in-segment diameter stenosis | 18.77 (14.43) | 22.82 (16.35)

41. Secondary Outcome: Target Vessel Failure (TVF)
Description: as for outcome 2
Time Frame: 5 years
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 605 | 286
percentage of participants | 20.3 | 26.6

42. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 9
Time Frame: 5 years
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 605 | 286
percentage of participants | 8.9 | 12.9

43. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: as for outcome 16
Time Frame: 5 years
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 605 | 286
percentage of participants | 8.8 | 11.9

44. Secondary Outcome: Ischemia Driven Major Adverse Cardiac Event (MACE)
Description: as for outcome 23
Time Frame: 5 years
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Number analyzed (Participants) | 605 | 286
percentage of participants | 14.4 | 22.0

ADVERSE EVENTS:
Arm/Group | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Serious Adverse Events (participants affected / at risk) | 219 | 126
Other Adverse Events (participants affected / at risk) | 71 | 55
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Abdominal pain (Gastrointestinal disorders) | 4/438 (4) | 3/211 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0/438 (0) | 1/211 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1/438 (1) | 0/211 (0)
Abscess limb (Infections and infestations) | 1/438 (1) | 0/211 (0)
Acute coronary syndrome (Cardiac disorders) | 2/438 (2) | 0/211 (0)
Acute myocardial infarction (Cardiac disorders) | 1/438 (1) | 1/211 (1)
Acute psychosis (Psychiatric disorders) | 0/438 (0) | 1/211 (1)
Adverse drug reaction (General disorders) | 0/438 (0) | 2/211 (2)
Agitation (Psychiatric disorders) | 0/438 (0) | 1/211 (1)
Anaemia (Blood and lymphatic system disorders) | 1/438 (3) | 5/211 (6)
Angina pectoris (Cardiac disorders) | 42/438 (51) | 37/211 (41)
Angina unstable (Cardiac disorders) | 4/438 (4) | 2/211 (2)
Anxiety (Psychiatric disorders) | 0/438 (0) | 1/211 (1)
Aortic aneurysm (Vascular disorders) | 1/438 (1) | 0/211 (0)
Aortic aneurysm repair (Surgical and medical procedures) | 1/438 (1) | 0/211 (0)
Aortic valve replacement (Surgical and medical procedures) | 1/438 (1) | 0/211 (0)
Appendicitis perforated (Gastrointestinal disorders) | 0/438 (0) | 1/211 (1)
Arrhythmia (Cardiac disorders) | 6/438 (7) | 2/211 (4)
Arterial thrombosis limb (Vascular disorders) | 1/438 (1) | 0/211 (0)
Arteriogram coronary (Investigations) | 2/438 (2) | 2/211 (2)
Arteriospasm coronary (Cardiac disorders) | 0/438 (0) | 1/211 (1)
Atherectomy (Surgical and medical procedures) | 3/438 (3) | 2/211 (2)
Atrial fibrillation (Cardiac disorders) | 2/438 (2) | 3/211 (3)
Atrial flutter (Cardiac disorders) | 0/438 (0) | 1/211 (1)
Atrioventricular block first degree (Cardiac disorders) | 1/438 (1) | 1/211 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0/438 (0) | 1/211 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/438 (1) | 0/211 (0)
Blood creatinine increased (Investigations) | 0/438 (0) | 2/211 (2)
Blood glucose increased (Investigations) | 3/438 (3) | 0/211 (0)
Blood pressure decreased (Investigations) | 1/438 (1) | 0/211 (0)
Body temperature increased (Investigations) | 1/438 (1) | 0/211 (0)
Bradycardia (Cardiac disorders) | 2/438 (2) | 2/211 (2)
Brain contusion (Injury, poisoning and procedural complications) | 0/438 (0) | 1/211 (1)
Breast lump removal (Surgical and medical procedures) | 1/438 (1) | 0/211 (0)
Cardiac enzymes increased (Investigations) | 0/438 (0) | 2/211 (2)
Cardiac failure congestive (Cardiac disorders) | 6/438 (8) | 6/211 (7)
Cardiac pacemaker replacement (Surgical and medical procedures) | 2/438 (2) | 0/211 (0)
Cardiac stress test abnormal (Investigations) | 2/438 (2) | 1/211 (1)
Cardiorespiratory arrest (Cardiac disorders) | 1/438 (1) | 0/211 (0)
Carotid artery stenosis (Nervous system disorders) | 2/438 (2) | 2/211 (2)
Carotid artery stent insertion (Surgical and medical procedures) | 1/438 (1) | 1/211 (1)
Carotid endarterectomy (Surgical and medical procedures) | 2/438 (2) | 0/211 (0)
Catheter site haematoma (General disorders) | 3/438 (3) | 2/211 (2)
Catheter site haemorrhage (General disorders) | 0/438 (0) | 1/211 (1)
Cellulitis (Infections and infestations) | 0/438 (0) | 1/211 (1)
Central nervous system lesion (Nervous system disorders) | 1/438 (1) | 0/211 (0)
Cerebrovascular accident (Nervous system disorders) | 4/438 (4) | 1/211 (2)
Cervicobrachial syndrome (Nervous system disorders) | 1/438 (1) | 0/211 (0)
Chest discomfort (General disorders) | 2/438 (2) | 3/211 (3)
Chest pain (Cardiac disorders) | 5/438 (5) | 1/211 (1)
Cholecystectomy (Surgical and medical procedures) | 1/438 (1) | 0/211 (0)
Cholecystitis (Hepatobiliary disorders) | 1/438 (1) | 1/211 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1/438 (1) | 0/211 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2/438 (3) | 1/211 (1)
Colectomy (Surgical and medical procedures) | 1/438 (1) | 1/211 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/438 (1) | 0/211 (0)
Colonic obstruction (Gastrointestinal disorders) | 1/438 (1) | 0/211 (0)
Colonic polyp (Gastrointestinal disorders) | 0/438 (0) | 1/211 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1/438 (1) | 0/211 (0)
Contusion (Injury, poisoning and procedural complications) | 1/438 (1) | 0/211 (0)
Cor pulmonale (Cardiac disorders) | 0/438 (0) | 1/211 (1)
Coronary angioplasty (Surgical and medical procedures) | 9/438 (9) | 9/211 (10)
Coronary arterial stent insertion (Surgical and medical procedures) | 3/438 (3) | 2/211 (2)
Coronary artery bypass graft (Surgical and medical procedures) | 10/438 (28) | 3/211 (5)
Coronary artery disease (Cardiac disorders) | 7/438 (7) | 0/211 (0)
Coronary artery dissection (Cardiac disorders) | 1/438 (1) | 1/211 (1)
Coronary artery occlusion (Cardiac disorders) | 2/438 (2) | 1/211 (1)
Coronary artery stenosis (Cardiac disorders) | 7/438 (7) | 3/211 (3)
Coronary artery thrombosis (Cardiac disorders) | 0/438 (0) | 1/211 (1)
Coronary revascularisation (Surgical and medical procedures) | 60/438 (94) | 43/211 (68)
Cough (Respiratory, thoracic and mediastinal disorders) | 1/438 (1) | 0/211 (0)
Deep vein thrombosis (Vascular disorders) | 0/438 (0) | 1/211 (1)
Dehydration (Investigations) | 1/438 (1) | 0/211 (0)
Dementia (Nervous system disorders) | 0/438 (0) | 1/211 (1)
Depression (Psychiatric disorders) | 0/438 (0) | 1/211 (1)
Device dislocation (Injury, poisoning and procedural complications) | 1/438 (1) | 0/211 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1/438 (1) | 0/211 (0)
Diarrhoea (Gastrointestinal disorders) | 2/438 (2) | 1/211 (1)
Diastolic dysfunction (Cardiac disorders) | 0/438 (0) | 1/211 (1)
Diverticulitis (Infections and infestations) | 2/438 (2) | 1/211 (1)
Dizziness (Nervous system disorders) | 4/438 (4) | 0/211 (0)
Dyspepsia (Gastrointestinal disorders) | 2/438 (2) | 0/211 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/438 (1) | 3/211 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1/438 (1) | 1/211 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1/438 (1) | 0/211 (0)
Electrocardiogram abnormal (Investigations) | 0/438 (0) | 1/211 (1)
Encephalopathy (Nervous system disorders) | 0/438 (0) | 1/211 (1)
Fall (Injury, poisoning and procedural complications) | 3/438 (3) | 1/211 (1)
Fatigue (General disorders) | 1/438 (1) | 0/211 (0)
Femoral arterial stenosis (Vascular disorders) | 1/438 (1) | 0/211 (0)
Fluid retention (Metabolism and nutrition disorders) | 1/438 (1) | 0/211 (0)
Fracture (Injury, poisoning and procedural complications) | 0/438 (0) | 1/211 (1)
Gallbladder disorder (Hepatobiliary disorders) | 1/438 (1) | 1/211 (1)
Gastric ulcer (Gastrointestinal disorders) | 1/438 (1) | 1/211 (1)
Gastritis erosive (Gastrointestinal disorders) | 0/438 (0) | 1/211 (1)
Gastroenteritis (Gastrointestinal disorders) | 0/438 (0) | 1/211 (1)
Gastroenteritis viral (Infections and infestations) | 0/438 (0) | 1/211 (1)
Gastrointestinal haemorrhage (Vascular disorders) | 6/438 (6) | 4/211 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0/438 (0) | 2/211 (2)
Gout (Metabolism and nutrition disorders) | 1/438 (1) | 0/211 (0)
Haemoglobin decreased (Investigations) | 1/438 (1) | 0/211 (0)
Headache (Nervous system disorders) | 1/438 (1) | 1/211 (1)
Hernia obstructive (General disorders) | 0/438 (0) | 1/211 (1)
Hiatus hernia (Gastrointestinal disorders) | 1/438 (1) | 0/211 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0/438 (0) | 1/211 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1/438 (1) | 0/211 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0/438 (0) | 1/211 (1)
Hypertension (Vascular disorders) | 1/438 (1) | 3/211 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0/438 (0) | 2/211 (2)
Hypotension (Vascular disorders) | 4/438 (4) | 2/211 (2)
Iliact artery stenosis (Vascular disorders) | 1/438 (1) | 0/211 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0/438 (0) | 1/211 (1)
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 0/438 (0) | 1/211 (1)
Implantable defibrillator replacement (Surgical and medical procedures) | 1/438 (1) | 0/211 (0)
Injury (Injury, poisoning and procedural complications) | 0/438 (0) | 1/211 (1)
Instent coronary artery restenosis (Cardiac disorders) | 1/438 (1) | 1/211 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0/438 (0) | 1/211 (1)
Knee arthroplasty (Surgical and medical procedures) | 1/438 (1) | 1/211 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0/438 (0) | 1/211 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/438 (0) | 1/211 (1)
Mitral valve incompetence (Cardiac disorders) | 1/438 (1) | 0/211 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0/438 (0) | 1/211 (1)
Myocardial infarction (Cardiac disorders) | 11/438 (11) | 10/211 (10)
Myocardial ischaemia (Cardiac disorders) | 25/438 (27) | 12/211 (15)
Nausea (Gastrointestinal disorders) | 0/438 (0) | 1/211 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/438 (1) | 0/211 (0)
Noncardiac chest pain (General disorders) | 16/438 (20) | 11/211 (14)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/438 (2) | 0/211 (0)
Operative haemorrhage (Injury, poisoning and procedural complications) | 1/438 (1) | 0/211 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/438 (0) | 1/211 (1)
Osteomyelitis (Infections and infestations) | 1/438 (1) | 0/211 (0)
Overdose (Injury, poisoning and procedural complications) | 0/438 (0) | 1/211 (1)
Pain (General disorders) | 1/438 (1) | 0/211 (0)
Pancreatitis (Gastrointestinal disorders) | 2/438 (2) | 0/211 (0)
Peripheral ischaemia (Vascular disorders) | 4/438 (4) | 3/211 (3)
Peripheral vascular disorder (Vascular disorders) | 1/438 (1) | 3/211 (3)
Phlebitis superficial (Vascular disorders) | 0/438 (0) | 1/211 (1)
Physical disability (Social circumstances) | 0/438 (0) | 1/211 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1/438 (1) | 0/211 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1/438 (1) | 0/211 (0)
Pneumonia (Infections and infestations) | 6/438 (6) | 1/211 (1)
Pneumonia fungal (Infections and infestations) | 1/438 (1) | 0/211 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/438 (1) | 0/211 (0)
Prostatectomy (Surgical and medical procedures) | 1/438 (1) | 0/211 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0/438 (0) | 1/211 (1)
Pyrexia (Gastrointestinal disorders) | 1/438 (1) | 0/211 (0)
Renal artery stenosis (Renal and urinary disorders) | 1/438 (1) | 0/211 (0)
Renal artery stent placement (Surgical and medical procedures) | 1/438 (1) | 1/211 (1)
Renal disorder (Renal and urinary disorders) | 0/438 (0) | 1/211 (1)
Renal failure (Renal and urinary disorders) | 1/438 (1) | 2/211 (4)
Renal failure acute (Renal and urinary disorders) | 1/438 (1) | 1/211 (1)
Renal failure chronic (Renal and urinary disorders) | 0/438 (0) | 1/211 (4)
Respiratory tract infection (Infections and infestations) | 0/438 (0) | 1/211 (1)
Retroperitoneal haemorrhage (Vascular disorders) | 2/438 (2) | 0/211 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1/438 (1) | 0/211 (0)
Sick sinus syndrome (Cardiac disorders) | 1/438 (1) | 0/211 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1/438 (1) | 0/211 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1/438 (1) | 0/211 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1/438 (1) | 1/211 (1)
Spinal operation (Surgical and medical procedures) | 1/438 (1) | 2/211 (2)
Staphylococcal infection (Infections and infestations) | 1/438 (1) | 0/211 (0)
Supraventricular tachycardia (Cardiac disorders) | 0/438 (0) | 1/211 (2)
Syncope (Nervous system disorders) | 5/438 (6) | 2/211 (2)
Tachycardia (Cardiac disorders) | 0/438 (0) | 1/211 (1)
Tachycardia paroxysmal (Cardiac disorders) | 1/438 (1) | 0/211 (0)
Thrombectomy (Surgical and medical procedures) | 1/438 (1) | 0/211 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1/438 (2) | 0/211 (0)
Thrombosis in device (Injury, poisoning and procedural complications) | 1/438 (1) | 0/211 (0)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/438 (0) | 1/211 (1)
Thyroidectomy (Surgical and medical procedures) | 1/438 (1) | 0/211 (0)
Transient ischaemic attack (Nervous system disorders) | 3/438 (3) | 1/211 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1/438 (1) | 0/211 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1/438 (1) | 0/211 (0)
Urinary retention (Renal and urinary disorders) | 0/438 (0) | 2/211 (2)
Urinary tract infection (Infections and infestations) | 1/438 (1) | 0/211 (0)
Urosepsis (Infections and infestations) | 0/438 (0) | 1/211 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1/438 (1) | 0/211 (0)
Vascular pseudoaneurysm (Vascular disorders) | 5/438 (5) | 3/211 (3)
Ventricular fibrillation (Cardiac disorders) | 1/438 (1) | 0/211 (0)
Ventricular tachycardia (Cardiac disorders) | 0/438 (0) | 1/211 (1)
Vertigo (Ear and labyrinth disorders) | 1/438 (1) | 0/211 (0)
Vomiting (Gastrointestinal disorders) | 1/438 (1) | 2/211 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | XIENCE V® EECSS | TAXUS® EXPRESS2™ ECSS
Angina pectoris (Cardiac disorders) | 71/438 (93) | 35/211 (44)
Catheter site haematoma (General disorders) | 12/438 (12) | 11/211 (11)
Myocardial infarction (Cardiac disorders) | 7/438 (7) | 11/211 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No